CLINICAL TRIAL: NCT00378066
Title: A Phase II Study of Combination Chemotherapy With Bevacizumab, Capecitabine and Oxaliplatin in Patients With Previously Untreated Metastatic or Recurrent Colorectal Cancer
Brief Title: Phase II Study of Bevacizumab, Capecitabine and Oxaliplatin in Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-ONCGI-0277
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Active Comparator): Bevacizumab, capecitabine and oxaliplatin for metastatic colorectal cancer, 1st line treatment
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab, Capecitabine, Oxaliplatin
  Other Names: Capecitabine, Oxaliplatin

SUMMARY:
The purpose of this study is to determine the efficacy and safety of bevacizumab/capecitabine/oxaliplatin combination in metastatic or recurrent Korean colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented colorectal adenocarcinoma
* ECOG performance status of 2 or lower
* Adequate bone marrow function
* Adequate kidney function
* Adequate liver function
* Informed consent

Exclusion Criteria:

* Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start
* Known allergy to study drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-08; Primary Completion 2006-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
time to progression | 6 months

SECONDARY OUTCOMES:
overall survival, safety, response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, M.D., Principal Investigator — Asan Medical Center
Locations (6):
- South Korea (6):
  - National Cancer Center, Goyang
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Hospital, Seoul
  - Bundang Seoul National University Hospital, Sungnam